CLINICAL TRIAL: NCT01920074
Title: A Phase 4, Multiple-dose, Pharmacokinetic, Safety, and Exploratory Efficacy Study of Nitroglycerin Ointment 0.4% (RECTIV®) in Adolescents (Age ≥12 to <17 Years) With Moderate to Severe Pain Due to Chronic Anal Fissure
Brief Title: Pharmacokinetic,Safety and Exploratory Efficacy of RECTIV® in Adolescents With Chronic Anal Fissure
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to study enrollment challenges that impacted the feasibility of conducting the study.
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APT-NIT_S-PRO-M_PEDKPK1_E
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Anal Fissure
Keywords: Anal Fissure; Nitroglycerin; Pediatrics; RECTIV®; Pediatric Research Equity Act
MeSH Terms: conditions — Fissure in Ano

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rectiv (Experimental)
  Interventions: Drug: Nitroglycerin Ointment 0.4%

INTERVENTIONS:
Drug: Nitroglycerin Ointment 0.4%

SUMMARY:
RECTIV® is an ointment containing 0.4% nitroglycerin (NTG) for the treatment of moderate to severe pain associated with chronic anal fissure approved in June 2011 by the US Food and Drug Administration (FDA) for adults. The purpose of this study is to assess the safety, pharmacokinetics, and exploratory efficacy of RECTIV® in adolescents

DETAILED DESCRIPTION:
This is an open-label, multicenter study conducted in up to 10 sites in the United States. A total of 13 pediatric male or female patients age ≥12 to <17 years will be enrolled. The patients will administer a dose of Rectiv® twice daily to characterize the safety, pharmacokinetics , and exploratory efficacy of Nitroglycerin Ointment 0.4% (RECTIV® )over 5 days

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥12 and <17 years of age
* At least 1 anal fissure for a minimum of 3 weeks in duration
* Anal fissure pain experienced over the last 24 hours at Screening and before enrollment
* Patient (and parent or caregiver as appropriate) has provided written informed consent

Key Exclusion Criteria:

* Current diagnosis of hemorrhoids
* Hypersensitivity, allergy, or contraindication to nitroglycerin
* History of hypertension and/or cardiovascular disease
* History or current diagnosis of inflammatory bowel disease
* History or current diagnosis of fistula(e)-in-ano or an anal abscess
* Fibrotic anal stenosis
* Previous anal surgery
* Diagnosis of cancer
* History of migraine or chronic headaches requiring treatment with analgesics
* Pregnant or lactating female patients
* Weight <36 kg

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Noncompartmental pharmacokinetic (PK) analyses will be performed on the full pharmacokinetic curves for NTG and its metabolites (1,2 glyceryl dinitrate and 1,3 glyceryl dinitrate) on Day 5 | Day 5
  The following PK parameters will be calculated as data permit:
  * Maximum observed concentration (Cmax)
  * Time of the maximum observed plasma concentration (Tmax)
  * Area under the concentration time curve from dosing up to the last quantifiable concentration (AUC0-last).
  * Area under the concentration time curve from dosing up to 480 minutes (AUC0-480)
  * The extrapolated area under the concentration time curve from dosing up to 12 hours (AUC0-12h) also will be calculated if quantifiable concentrations are observed during the entire dose interval.
  * Terminal elimination half-life (t1/2) On the basis of the results of the study, additional noncompartmental PK parameters may be calculated and reported.
  In addition, a population PK model for NTG will be developed based on the PK data from Day 5. By using this model, the following additional PK parameters may be reported:
  * Apparent volume of distribution (V/F)
  * Apparent clearance (CL/F)

SECONDARY OUTCOMES:
• Absolute change from baseline in 24-hour average anal fissure pain scores assessed by the Wong-Baker FACES® and the Numerical Rating Scale for pain after each evening dose over days 1 through 4 | Day 5

OTHER OUTCOMES:
To assess the safety of Rectiv® in adolescents (age ≥12 to <17 years) | Screening through the completion of study participation
  Safety and tolerability are assessed through adverse events (AEs), clinical laboratory test results (hematology, serum biochemistry, and urinalysis), vital sign measurements (heart rate, supine and orthostatic blood pressure, oral temperature, and respiratory rate), 12-lead ECG results, anal area assessment, physical examination findings (including body weight), and concomitant medications (including the use of rescue acetaminophen for headaches).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hyman, MD, Principal Investigator — Children's Hospital New Orleans, LA; Taryn Weissman, MD, Study Director
Locations (6):
- United States (6):
  - Children's Hospital, Los Angeles, California
  - Advanced Medical Research Center, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Willis-Knighton Pediatric GI Specialist, Shreveport, Louisiana
  - Children's Mercy Hospital, Kansas City, Missouri
  - Sealy Urgent Care Center and Medical Clinic, Sealy, Texas

REFERENCES:
- [Result] Demirbag S, Tander B, Atabek C, Surer I, Ozturk H, Cetinkursun S. Long-term results of topical glyceryl trinitrate ointment in children with anal fissure. Ann Trop Paediatr. 2005 Jun;25(2):135-7. doi: 10.1179/146532805X45737. PMID 15949202
- [Result] Kenny SE, Irvine T, Driver CP, Nunn AT, Losty PD, Jones MO, Turnock RR, Lamont GL, Lloyd DA. Double blind randomised controlled trial of topical glyceryl trinitrate in anal fissure. Arch Dis Child. 2001 Nov;85(5):404-7. doi: 10.1136/adc.85.5.404. PMID 11668104
- [Result] Schiano di Visconte M, Di Bella R, Munegato G. Randomized, prospective trial comparing 0.25 percent glycerin trinitrate ointment and anal cryothermal dilators only with 0.25 percent glycerin trinitrate ointment and only with anal cryothermal dilators in the treatment of chronic anal fissure: a two-year follow-up. Dis Colon Rectum. 2006 Dec;49(12):1822-30. doi: 10.1007/s10350-006-0731-y. PMID 17096178